CLINICAL TRIAL: NCT03275467
Title: Faecal Microbiota Transplantation in Patients With Microscopic Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Region Örebro County (Other)
Responsible Party: Principal Investigator, Robert Brummer, Professor, Örebro University, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/072
Record Dates: First submitted 2017-08-28; First posted 2017-09-07 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Faecal microbiota transfer (FMT) (Experimental): Suspended stool from a healthy donor
  Interventions: Other: Faecal microbiota transfer (FMT)

INTERVENTIONS:
Other: Faecal microbiota transfer (FMT) — Suspended stool from a healthy donor

SUMMARY:
Microscopic colitis (MC) is a disease with chronic inflammation of the colon that is mostly diagnosed in middle-aged or elderly women. Patients suffer from chronic watery diarrhoea, abdominal pain and weight loss. The aetiology of MC is still unknown but it is hypothesized that MC is caused by a deregulated immune response to a luminal agent in predisposed individuals, and an important role of the intestinal microbiota is suggested.

In the current proof-of-concept study, the effect of faecal microbiota transfer (FMT) in 10 MC patients will be evaluated. FMT consists in the infusion of suspended stool from a healthy donor into the intestine of a patient with the aim to restore a disturbed intestinal microbiota.

DETAILED DESCRIPTION:
This will be an intervention pilot study with a 12-week and an optional 6-months follow-up period. It will be investigated if the infusion of suspended stool from healthy donors improves the symptoms of MC patients by restoring their disturbed intestinal microbiota. This procedure is known as faecal microbiota transplantation (FMT).

MC patients (n=10) will be randomised to receive FMT using stool from one of two healthy donors.

At baseline, blood samples and mucosal biopsies will be obtained from the descending colon. In addition, faecal samples will be collected and patients will complete symptom questionnaires. The first FMT will be administered by colonoscopy, FMT 2-3 by enemas. Faecal samples will be collected and questionnaires will be completed at different time points during the study. The patients will be followed-up at 6 weeks, 8 weeks, 12 weeks and 6 months after receiving FMT 1, however, the follow-up after 6 months will be optional. Additional biopsies from the descending colon and blood samples will be collected 6 weeks after the first FMT.

ELIGIBILITY:
Inclusion criteria for patients:

1. Signed informed consent
2. Active MC diagnosis, defined as >3 stools a day from which at least one should be watery
3. Willingness to stop budesonide treatment during participation in the trial
4. Age: 18-70 years

Exclusion criteria for patients

1. Previous complicated gastrointestinal surgery
2. Malignant disease except non-melanoma skin cancer
3. Dementia, severe depression, major psychiatric disorder, or other incapacity for adequate cooperation
4. C. difficile or other current gastroenteritis
5. Females who are pregnant or breast-feeding
6. Severe endometriosis
7. Antimicrobial treatment 4 weeks prior to first screening visit
8. Antimicrobial prophylaxis (eg. acne, urinary tract infection)
9. Regular consumption of probiotic products 4 weeks prior to randomization
10. Recently diagnosed lactose intolerance (less than 6 months prior to first screening visit)
11. Recently diagnosed coeliac disease (less than 6 months prior to first screening visit)
12. Regular intake of NSAIDs (non steroidal anti-inflammatory drugs)
13. Abuse of alcohol or drugs
14. Any clinically significant disease/condition which in the investigator's opinion could interfere with the results of the trial

Inclusion criteria for donors

1. Signed informed consent
2. High-butyrate producing microbiota in faecal samples
3. Age: 18-65 years

Exclusion criteria for donors

1. Known organic gastrointestinal disease (e.g. IBD, IBS, chronic diarrhoea or constipation)
2. First degree relative with IBD
3. History of or present gastrointestinal malignancy or polyposis
4. Recent (gastrointestinal) infection (within last 6 months)
5. History of major gastrointestinal surgery (e.g. gastric bypass)
6. Eosinophilic disorders of the gastrointestinal tract
7. Current communicable disease (e.g. upper respiratory tract infection)
8. Malignant disease and/or patients who are receiving systemic anti-neoplastic agents
9. Psychiatric diseases (e.g. dementia, depression, schizophrenia, autism, Asperger Syndrome) or other incapacity for adequate cooperation
10. Chronic neurological/neurodegenerative diseases (e.g. Parkinson's disease, multiple sclerosis)
11. Autoimmune disease and/or patients receiving immunosuppressive medications
12. Major relevant allergies (e.g. food allergy, multiple allergies)
13. Chronic pain syndromes (e.g. fibromyalgia)
14. Chronic fatigue syndrome
15. HIV, hepatitis A, B, C or known exposure within the recent 12 months
16. Obesity (BMI>30) or metabolic syndrome
17. Antimicrobial treatment or prophylaxis within the last 3 months
18. Other chronic use of drugs that may affect the microbiome, e.g. proton pump inhibitors
19. First degree relative with cardiovascular thrombosis before 50 years of age
20. Females who are pregnant or breast-feeding
21. Known clinically significant abnormal laboratory values
22. Participation in high-risk sexual behaviours
23. Abuse of alcohol or drugs
24. Tattoo or body piercing within the last 6 months
25. Travelling in countries with low hygiene or high infection risk for endemic diarrhoea within the last 6 months
26. Positive stool testing for C. difficile, ova and parasites (e.g. Cyclospora, Isospora, Cryptosporidium), enteric pathogens (e.g. enterohaemorrhagic E. coli, Salmonella, Shigella, Yersinia, Campylobacter, Giarda antigen, amoebas)
27. Positive stool testing for multiresistant bacteria (e.g. extended-spectrum beta- lactamase (ESBL) producing organisms, multi-resistant Gram-negative bacilli (MRGN) 3 and 4, vancomycin-resistant enterococci (VRE) or methicillin-resistant Staphylococcus aureus (MRSA))
28. Calprotectin > 50 μg/g of faeces
29. Positive blood testing for HIV, Hepatitis A, B, C, syphilis, Human T-lymphotropic virus (HTLV), cytomegalovirus (CMV) and Epstein Barr Virus (EBV)
30. Any clinically significant disease/condition which in the investigator's opinion could interfere with the results of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of MC patients in remission six weeks after the first FMT. | 6 weeks
  Remission is defined as <3 stools per day and a mean of less than one watery stool per day.

SECONDARY OUTCOMES:
Changes in general health and symptom questionnaire scores | 6 weeks, 8 weeks, 12 weeks, 6 months
  SHS
Changes in general health questionnaire scores | 6 weeks, 8 weeks, 12 weeks, 6 months
  SF-36
Changes in quality of life questionnaire scores | 6 weeks, 8 weeks, 12 weeks, 6 months
  EG-5D-5L
Changes in gastrointestinal symptom questionnaire scores | 6 weeks, 8 weeks, 12 weeks, 6 months
  GSRS
Changes in hospital and anxiety depression scores | 6 weeks, 8 weeks, 12 weeks, 6 months
  HADS
Changes in number and form of bowel movements | 6 weeks, 8 weeks, 12 weeks, 6 months
  1-week-diaries
Changes in faecal and mucosal microbiota composition | faecal: 6 weeks, 8 weeks, 12 weeks, 6 months; mucosal: 6 weeks
  16S rRNA-based next generation sequencing
Changes in lymphocyte infiltration | 6 weeks
  Immunohistochemistry and flow cytometry
Changes in subepithelial collagen layer | 6 weeks
  Immunohistochemistry
Changes in immune cell composition of colonic biopsies | 6 weeks
  Immunohistochemistry and flow cytometry

OTHER OUTCOMES:
Changes in inflammation markers in faecal samples such as faecal calprotectin | 6 weeks, 8 weeks, 12 weeks, 6 months
Changes in metabolite profile in faecal samples and blood | faecal: 6 weeks, 8 weeks, 12 weeks, 6 months; blood: 6 weeks
Changes in gene expression in mucosal biopsies | 6 weeks
Changes in barrier function markers in colonic biopsies | 6 weeks
Changes in gene expression of butyrate transporters in colonic biopsies | 6 weeks
Changes in markers of inflammation and intestinal barrier function in blood | 6 weeks
Changes in plasma levels of cardiovascular disease markers and platelet responsiveness and aggregation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, Professor, MD, Principal Investigator — Örebro University, Sweden
Locations (1):
- University Hospital Örebro, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No